CLINICAL TRIAL: NCT00753103
Title: Phase II Pilot Cohort Study to Investigate the Safety and Efficacy of Infliximab as Additional Therapy in the Treatment if Anti-Neutrophil Cytoplasm Antibody Associated Vasculitis
Brief Title: Anti-Cytokine Therapy for Vasculitis
Acronym: ACTIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Dr Lorraine Harper, University Hospitals Birmingham NHS Foundation Trust/University of Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRK2031
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Wegener's Granulomatosis; Renal Limited Vasculitis; Microscopic Polyangiitis
Keywords: Infliximab; Vasculitis; antitnf monoclonal antibody
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Vasculitis | interventions — Infliximab; Cyclophosphamide; Prednisolone; Azathioprine; Plasma Exchange; Mycophenolic Acid; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients with active vasculitis who receive infliximab in addition to standard immunosuppressive therapy
  Interventions: Biological: Infliximab; Drug: Cyclophosphamide; Drug: Prednisolone; Drug: Azathioprine; Drug: Mycophenolate mofetil; Drug: Methylprednisolone
- 2 (Active Comparator): Patients with active ANCA associated vasculitis who receive standard immunosuppression but no infliximab
  Interventions: Drug: Cyclophosphamide; Drug: Prednisolone; Drug: Azathioprine; Procedure: Plasma exchange; Drug: Mycophenolate mofetil; Drug: Methylprednisolone

INTERVENTIONS:
Biological: Infliximab — 5 mg/kg intravenous infusion at weeks 0, 2, 6 and 10 of study
  Other Names: Remicade
  Arms: 1
Drug: Cyclophosphamide — Daily oral 2 mg/kg or pulsed intravenous 15mg/kg every 2-3 weeks for 3-6 months (until patient has been in remission for 3 months).
Drug: Prednisolone — Daily oral 1mg/kg tapered over 12 months
Drug: Azathioprine — Daily oral 2 mg/kg started once patient is in remission and cyclophosphamide has been discontinued.
Procedure: Plasma exchange — Additional therapy for patients with severe vasculitis (creatinine > 500 mcmol/L or pulmonary haemorrhage). 7x 4L exchanges over 10 days.
  Arms: 2
Drug: Mycophenolate mofetil — Daily oral up to 1.5 g twice daily as tolerated. Used as alternative to azathioprine at lead physicians discretion.
Drug: Methylprednisolone — 500 mg intravenous infusion daily for three days at lead physicians discretion.

SUMMARY:
The purpose of this study is to determine whether Infliximab (monoclonal anti-tumour necrosis factor alpha antibodies) are safe and effective in the treatment of anti-neutrophil cytoplasm antibody (ANCA) associated vasculitis.

DETAILED DESCRIPTION:
Anti-neutrophil cytoplasm antibody (ANCA) associated vasculitis is a life-threatening systemic inflammatory autoimmune disease. Current treatment regimes using corticosteroids and cyclophosphamide have improved patient survival but are associated with treatment associated morbidity and mortality. Tumour necrosis factor alpha (TNF) is a proinflammatory cytokine which has been implicated in the pathogenesis of ANCA vasculitis. Anti-TNF therapies have been used successfully in the management of other inflammatory autoimmune diseases. This phase II cohort study has been designed to investigate the safety and efficacy of anti-TNF monoclonal antibody (Infliximab) therapy for patients with ANCA associated vasculitis when used in addition to standard immunosuppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Either newly diagnosed or relapsed ANCA associated vasculitis (Wegener's granulomatosis, microscopic polyangiitis, renal limited vasculitis)

Exclusion Criteria:

* Active infection
* Malignancy
* Pregnancy
* Diagnosis of Churg-Strauss syndrome or anti-glomerular basement membrane antibody disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2003-01; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Time to clinical remission (Birmingham Vasculitis Activity Score 0 or 1) | 0, 6, 10, 14, 26, 39 and 52 weeks

SECONDARY OUTCOMES:
Adverse events | Weeks 2, 6, 10, 14, 26, 39, 52
Vasculitis Damage Index Score | Weeks 0, 14, 26, 39, 52
Renal function | Weeks 0, 2, 6, 10, 14, 26, 39, 52

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Harper, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom